CLINICAL TRIAL: NCT04732559
Title: General Attitudes Towards Surrogacy in Poland
Status: Completed | Type: Observational
Sponsor: University of Gdansk (Other)
Collaborators: Principal Investigator: Karolina Lutkiewicz, PhD (Unknown); Sub-Investigator: Łucja Bieleninik, PhD (Unknown); Sub-Investigator: Mariola Bidzan, Prof (Unknown)
Responsible Party: Principal Investigator, Karolina Lutkiewicz, PhD, Assistant Professor, University of Gdansk
Other Study IDs: 46/2020
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Surrogate Mothers
Keywords: traditional surrogacy; gestational surrogacy; attitudes; surrogate parenthood
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to:

- investigate the general attitudes towards surrogacy among Polish population.

The secondary aims of the study are as follows:

* assess the differences in attitudes towards traditional vs. gestational surrogacy among Polish population,
* assess the cognitive concerns about issues related to surrogacy,
* assess the acceptance of surrogate parenthood,
* assess the attitude towards the surrogate mother,
* identify factors that influence the attitudes towards surrogacy,
* examine if there are differences in attitudes among members of the general public, health care professionals, students (health/medical studies vs. non-medical studies) and people with infertility diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* no restrictions to gender
* age ≥ 18
* able to understand and complete the questionnaire in Polish
* country of residence: Poland

Exclusion Criteria:

• if at least one of the inclusion criteria is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population in Poland with the divison to subgroups to examine differences between attitudes towards surrogacy among men and women, medical staff/personnel, students of medical and health studies with students of other disciplines and people with diagnosed infertility.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
General attitudes towards surrogacy. | Through study completion, an average of 1 year
  Attitudes Towards Surrogacy Survey (ATSS) was constructed on the basis of a literature review and other existing questionnaires or surveys. The survey consists of 15 items. The opinion is indicated by using seven-point Likert-type scale (1= strongly disagree, 7= strongly agree). For most items a higher score indicates a more positive attitude towards surrogacy. To prevent acquiescence response bias, 4 items were reversed. Total score was obtained by summing the items, ranging from 15 (minimum negative attitude) to 105 (maximum positive attitude).

SECONDARY OUTCOMES:
Attitudes towards traditional vs. gestational surrogacy | Through study completion, an average of 1 year
  Measured by the Attitudes to Surrogate Parenthood Questionnaire (ASPQ) constructed by Constantinidis D., Roger Cook (2012). The opinion was indicated by using seven-point Likert-type scale (1= strongly disagree, 7= strongly agree). One item included yes/no answer.
The Cognitive Concerns About Issues Related to Surrogacy Scale (CCAIRSS) | Through study completion, an average of 1 year
  Measured by the Attitudes to Surrogate Parenthood Questionnaire (ASPQ) constructed by Constantinidis D., Roger Cook (2012). The Cognitive Concerns About Issues Related to Surrogacy Scale (CCAIRSS) was used in order to examine the level of concerns and different complications associated to traditional and gestational surrogacy. Participants use five-point Likert-type scale to express how much they agree with each statement. Total score was obtained by summing the items, ranging from 15 to 75. High scores reflected smaller surrogacy-related concers and low scores reflected greater surrogacy-related concerns (Constantinidis, Cook, 2012).
Attitudes towards the acceptance of surrogate parenthood | Through study completion, an average of 1 year
  Measured by the Attitudes to Surrogate Parenthood Questionnaire (ASPQ) constructed by Constantinidis D., Roger Cook (2012). The opinion was indicated by using five-point Likert-type scale (1= strongly disagree, 5= strongly agree). Some items included yes/no answer and ranking.
Attitudes towards the surrogate mother | Through study completion, an average of 1 year
  Measured by the Attitudes to Surrogate Parenthood Questionnaire (ASPQ) constructed by Constantinidis D., Roger Cook (2012). The opinion was indicated by using five-point Likert-type scale (1= strongly disagree, 5= strongly agree).
Socio-demographic factors | Through study completion, an average of 1 year
  Measured by the socio-demographic survey designed for the purpose of the study, which capture the following factors: gender, age, place of living, education background, work background, marital status, sexual orientation, religion and diagnosis of infertility.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available on request from the corresponding author. The data are not publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Background] Constantinidis D, Cook R. Australian perspectives on surrogacy: the influence of cognitions, psychological and demographic characteristics. Hum Reprod. 2012 Apr;27(4):1080-7. doi: 10.1093/humrep/der470. Epub 2012 Jan 30. PMID 22294557
- [Derived] Lutkiewicz K, Bieleninik L, Jurek P, Bidzan M. Attitudes towards surrogacy in the context of socio-demographic determinants: a cross-sectional study. J Reprod Infant Psychol. 2025 Jun 6:1-16. doi: 10.1080/02646838.2025.2513662. Online ahead of print. PMID 40474789